CLINICAL TRIAL: NCT06913452
Title: Effect of Obesity on Tear Film and Ocular Health Among Diabetic Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSRSW/Batch-Fall23/800
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Tear Film Deficiency
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the effect of obesity on tear film and ocular health in diabetic patients.

Research Design An observational cross-sectional study will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18+ years)
* diagnosed with type 1 or type 2 diabetes
* categorized as obese or non-obese (BMI >30 or <30)
* stable glycemic control, and willing to provide consent.

Exclusion Criteria:

* Non-diabetic individuals
* pregnant/lactating women
* those with recent ocular surgeries
* systemic medications affecting tear film, or severe unrelated diseases.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic participants aged 18-70 with varying BMI categories will be assessed for tear production and film stability using Schirmer's Test and Tear Break-Up Time (TBUT). Demographics, medical history, and ocular health will also be recorded in a controlled clinic environment.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
The Oswestry Disability Index (ODI) | 12 Months
  The Oswestry Disability Index (ODI) is a questionnaire used to assess functional disability in individuals with low back pain, with scores ranging from 0% (no disability) to 100% (maximum disability), and interpreted as follows: 0-20% minimal disability, 21-40% moderate, 41-60% severe, 61-80% crippling, and 81-100% bed-bound or exaggerated symptom

CONTACTS AND LOCATIONS:
Locations (1):
- Alvi Hospital, Mandi Bahāuddīn, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No